CLINICAL TRIAL: NCT02603562
Title: An Open-Label, Intrapatient Dose-Escalation Study to Evaluate the Safety, Tolerability, Immunogenicity, and Biological Activity of ATYR1940 in Patients With Early Onset and Other Pediatric Onset Facioscapulohumeral Muscular Dystrophy
Brief Title: Evaluate Safety and Biological Activity of ATYR1940 in Participants With Early Onset Facioscapulohumeral Muscular Dystrophy
Acronym: FSHD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: aTyr Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATYR1940-C-003; 2014-003346-27 (EudraCT Number)
Record Dates: First submitted 2015-11-05; First posted 2015-11-13 (Estimated); Results first posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-09

CONDITIONS: Facioscapulohumeral Muscular Dystrophy (FSHD)
Keywords: FSHD
MeSH Terms: conditions — Muscular Dystrophy, Facioscapulohumeral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ATYR1940 (Experimental): Participants received ATYR1940 intravenous (IV) infusion at doses of 0.3, 1.0, and 3.0 milligrams/kilograms (mg/kg) once weekly using intraparticipant dose escalation for 12 weeks.
  Interventions: Biological: ATYR1940

INTERVENTIONS:
Biological: ATYR1940 — Concentrate for solution for infusion

SUMMARY:
The purpose of this study is to assess the safety and biological activity of ATYR1940 in participants with early onset FSHD.

DETAILED DESCRIPTION:
A Phase 1b/2 open-label, intraparticipant dose-escalation study aiming to evaluate the safety, tolerability, immunogenicity, biological and pharmacodynamic activity of intravenous ATYR1940, administered once weekly for 12 weeks, in early onset FSHD participants with signs or symptoms prior to 10 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Established, genetically confirmed diagnosis of FSHD.
* Onset of FSHD signs or symptoms prior to 10 years of age, as documented in the participant's medical record or based on participant or family report.
* Provide written informed consent or assent
* In the Investigator's opinion, participant is willing and able to complete all study procedures and comply with the weekly study visit schedule.

Exclusion Criteria:

* Currently receiving treatment with an immunomodulatory agent including targeted biological therapies within the 3 months before baseline; corticosteroids within 3 months before baseline; or high-dose non-steroidal anti-inflammatory agents within 2 weeks before baseline.
* Currently receiving curcumin or albuterol; use of a product that putatively enhances muscle growth or activity on a chronic basis within 4 weeks before baseline; statin treatment initiation or significant adjustment to statin regimen within 3 months before baseline (stable, chronic statin use is permissible).
* Use of an investigational product or device within 30 days before baseline.
* Evidence of an alternative diagnosis other than FSHD or a coexisting myopathy or dystrophy, based on prior muscle biopsy or other available investigations.
* History of severe restrictive or obstructive lung disease, or evidence for interstitial lung disease on screening chest radiograph.
* History of anti-synthetase syndrome, prior Jo-1 Ab-positivity, or a positive or equivocally positive Jo-1 Ab test result during screening.
* Chronic infection, such as hepatitis B, hepatitis C, or human immunodeficiency virus or a history of tuberculosis.
* Vaccination within 8 weeks before baseline or vaccination is planned during study participation.
* Symptomatic cardiomyopathy or severe cardiac arrhythmia, that may, in the Investigator's opinion, limit the participant's ability to complete the study protocol.
* Muscle biopsy within 30 days before baseline.

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2016-03-30 (Actual); Primary Completion 2016-12-12 (Actual); Study Completion 2016-12-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (4):
  - Stanford University, Stanford, California
  - University of Iowa Children's Hospital, Iowa City, Iowa
  - OSU Wexner Medical Center, Columbus, Ohio
  - University of Utah, Salt Lake City, Utah
- France (2):
  - Centre d'nvestigation Clinique - Centre de Pharmacologie Clinique et d'Evaluations Thérapeutiques (CICCPCET), Marseille
  - Institut de Myologie, Paris
- Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta, Milan, Italy

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ATYR1940
Started | 8
Received at Least 1 Dose of Study Drug | 8
Completed | 7
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least 1 full or partial dose of ATYR1940 and had a post-infusion safety observation.
Groups:
- ATYR1940: Participants received ATYR1940 IV infusion at doses of 0.3, 1.0, and 3.0 mg/kg once weekly using intraparticipant dose escalation for 12 weeks.
Arm/Group | ATYR1940
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 17.9 [16 to 20]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: TEAEs were defined as adverse events (AEs) with an onset following administration of the first dose of study drug. AEs were defined as any untoward medical occurrence in a participant administered study drug and that does not necessarily have a causal relationship with the study drug. Worsening of a pre-existing medical condition should have been considered an AE if there was either an increase in severity, frequency, or duration of the condition or an association with significantly worse outcomes. SAEs were defined as any AE that, in the view of either the Investigator or Sponsor, resulted in any of the following outcomes as fatal, life-threatening, required in-participant hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, a congenital anomaly/birth defect, an important medical event. A summary of all SAEs and Other AEs (nonserious) regardless of causality is located in 'Reported Adverse Events' Section.
Time Frame: Up to End of Study (up to Week 25)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | ATYR1940
Number analyzed (Participants) | 8
Participants
  TEAEs | 8
  SAEs | 0

2. Primary Outcome: Number of Participants With a Clinical Laboratory Abnormality Leading to an AE
Description: Laboratory parameters included hematology (hematocrit, hemoglobin, red blood cell count, white blood cell count with differential [neutrophils, lymphocytes, monocytes, eosinophils, basophils], and platelet count); serum chemistries (blood urea nitrogen, creatinine, total bilirubin, aspartate aminotransferase, alanine aminotransferase, gamma-glutamyl transferase, alkaline phosphatase, total protein, sodium, potassium, bicarbonate, calcium, chloride, magnesium, inorganic phosphate, creatine kinase, lactate dehydrogenase, erythrocyte sedimentation rate, C-reactive protein, troponin, myoglobin, insulin-like growth factor 1, and cholesterol [nonfasting]); and urinalysis (color, pH, specific gravity, protein, glucose, ketones, and blood). Clinically significant laboratory abnormalities were based upon Investigator's discretion. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Up to End of Study (Up to Week 25)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | ATYR1940
Number analyzed (Participants) | 8
Participants | 1

3. Primary Outcome: Number of Participants With an Ocular Abnormality Leading to a TEAE
Description: Ocular parameters included vitreous, retina, macula, choroid, optic nerve, and optic nerve pallor. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Up to End of Study (Up to Week 25)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | ATYR1940
Number analyzed (Participants) | 8
Participants | 0

4. Primary Outcome: Number of Participants With an Impact on Hearing From ATYR1940 Treatment
Time Frame: Up to End of Study (Up to Week 25)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | ATYR1940
Number analyzed (Participants) | 8
Participants | 0

5. Primary Outcome: Number of Participants With a Clinically Significant Pulmonary Function Event Resulting in a TEAE
Description: Pulmonary evaluations included pulmonary function tests and pulse oximetry. Clinically significant changes were to be reported as adverse events. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Up to End of Study (up to Week 25)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | ATYR1940
Number analyzed (Participants) | 8
Participants | 0

6. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibodies (ADA)
Description: Titers through Week 12 are summarized.
Time Frame: Baseline up to Week 12
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | ATYR1940
Number analyzed (Participants) | 8
Participants | 4

7. Secondary Outcome: Number of Participants With a Jo-1 Antibody (Ab) Test Result ≥1.5 Units/Milliliter (U/mL)
Description: Participants with Jo-1 Ab levels ≥1.5 units/milliliter (U/mL) were to be discontinued from dosing of the study drug.
Time Frame: Baseline up to Week 12
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | ATYR1940
Number analyzed (Participants) | 8
Participants | 0

8. Secondary Outcome: Number of Participants With Infusion-Related Reactions
Description: Infusion-related reactions included fever, chills, rigors, myalgia, facial erythema, systemic erythema, pallor, facial swelling, chest tightness, difficulty breathing, wheezing, stridor, tachypnea, bronchospasm, cough, tachycardia, significant pulse rate increase from baseline without obvious cause, bradycardia, significant pulse rate decrease from baseline, pre-syncope or syncope, hypotension, orthostatic hypotension, blood pressure swings (including hypertension), skin rash, urticaria, angioedema, pruritus, difficulty speaking, hoarse voice, raspy voice, excessive salivation, difficulty swallowing, nausea, vomiting, cramps, diarrhea; swelling of the throat, tongue, mouth, or lip, and development of a headache especially moderate or greater after start of infusion. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Baseline up to Week 12
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | ATYR1940
Number analyzed (Participants) | 8
Participants | 1

9. Secondary Outcome: Percent Change From Baseline in Manual Muscle Testing (MMT) Score at Week 14
Description: MMT was graded on a scale from 0 (no movement) to 10 (normal movement). Each side of the body and the position in which each muscle was tested were recorded for each participant. The total MMT score were calculated by averaging a converted-MMT scores across all tested muscle groups. Decreased motor function was indicated by decreased individual muscle or composite MMT score.
Time Frame: Baseline, Week 14
Population: as for baseline characteristics
Measure: Mean (Full Range); unit: percent change
Arm/Group | ATYR1940
Number analyzed (Participants) | 8
percent change | 3.8 [-6 to 19]

ADVERSE EVENTS:
Time Frame: Up to End of Study (Up to Week 25)
Description: Safety analysis set included all participants who received at least 1 full or partial dose of ATYR1940 and had a post-infusion safety observation. Serious Adverse Event and Other Adverse Event data were prespecified to be collected as a single Arm/Group for any participant who received at least 1 dose of the study drug, regardless of their dose level.
Arm/Group | ATYR1940
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 8/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ATYR1940 (N=8)
Paraesthesia (Nervous system disorders) | 3
Headache (Nervous system disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Nasopharyngitis (Infections and infestations) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Ageusia (Nervous system disorders) | 1
Burning sensation (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Bronchitis (Infections and infestations) | 1
Conjunctivitis bacterial (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Post procedural contusion (Injury, poisoning and procedural complications) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Chills (General disorders) | 1
Pain (General disorders) | 1
Electrocardiogram P wave biphasic (Investigations) | 1
Troponin increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes